CLINICAL TRIAL: NCT00921557
Title: Impact of Oral Alendronate Therapy on Bone Mineral Density in HIV-infected Children and Adolescents With Low Bone Mineral Density
Brief Title: Safety and Effectiveness of Alendronate for Bone Mineral Density in HIV-infected Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P1076; 10669 (Registry Identifier: DAIDS-ES Registry Number); IMPAACT P1076
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2017-06

CONDITIONS: HIV Infection
Keywords: Bone mineral density
MeSH Terms: conditions — HIV Infections | interventions — Alendronate; Calcium Carbonate; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1A: Alendronate/Alendronate (Experimental): Participants received alendronate for 96 weeks and calcium carbonate/vitamin D for 144 weeks
  Interventions: Drug: Alendronate; Dietary Supplement: Calcium carbonate/vitamin D
- 1B: Alendronate/Placebo (Experimental): Participants received alendronate for 48 weeks followed by placebo for 48 weeks and calcium carbonate/vitamin D for 144 weeks
  Interventions: Drug: Alendronate; Drug: Placebo; Dietary Supplement: Calcium carbonate/vitamin D
- 2: Placebo/Alendronate (Experimental): Participants received placebo for 48 weeks followed by alendronate for 48 weeks and calcium carbonate/vitamin D for 144 weeks
  Interventions: Drug: Alendronate; Drug: Placebo; Dietary Supplement: Calcium carbonate/vitamin D

INTERVENTIONS:
Drug: Alendronate — Oral tablet taken once weekly: 70 mg if participant greater than 30 kg or 35 mg if participant less than or equal to 30 kg
  Other Names: Fosamax
Drug: Placebo — Oral tablet taken once weekly
  Arms: 1B: Alendronate/Placebo; 2: Placebo/Alendronate
Dietary Supplement: Calcium carbonate/vitamin D — Tablet taken once or twice daily: calcium carbonate (600 mg) and vitamin D (400 IU) once daily for participants with 25-OH-vitamin D levels greater than or equal to 20 ng/mL or twice daily for those with 25-OH-vitamin D levels less than 20 ng/mL

SUMMARY:
HIV-infected children, youth, and adults have lower bone mineral density (BMD) than would be expected for HIV-uninfected people of similar age, weight and race. As the majority of perinatally HIV-infected U.S. children are entering or in adolescence, the potential for HIV-related impaired BMD during the adolescent peak of bone mass acquisition is of particular concern. The primary purpose of this study was to compare changes from pre-treatment levels of BMD of the lumbar spine after 24 and 48 weeks of alendronate treatment with placebo in HIV-infected children and adolescents.

DETAILED DESCRIPTION:
Puberty is a time when the foundation is laid for healthy bone mass. Over the course of puberty, 26% of bone mass is established in the 4-year period of peak height velocity and up to 60% of adult peak bone mass is established. Factors that affect normal bone mineralization include calcium intake, vitamin D status, degree of physical and weight bearing activities, hormones, genetics, body weight, and general health and nutrition status. HIV-infected children, youth, and adults have lower bone mineral density (BMD) than would be expected for healthy people of similar age, weight, and race. As the majority of perinatally HIV-infected U.S. children are entering or in adolescence, the potential for HIV-related impaired BMD during the adolescent peak of bone mass acquisition is of particular concern. The purpose of this study was to compare changes in BMD of the lumbar spine from pre-treatment levels to 24 and 48 weeks after alendronate treatment or placebo in HIV-infected children and adolescents.

Participants were randomized equally into one of three groups: Group 1A received alendronate for 96 weeks; Group 1B received alendronate for 48 weeks followed by placebo for 48 weeks; Group 2 received placebo for 48 weeks followed by alendronate for 48 weeks. All three groups were followed off treatment for an additional 48 weeks. Participants also received vitamin D/calcium for the duration of the study and were asked to perform 60 minutes of weight-bearing exercise each day.

Clinic visits were scheduled every 12 weeks after entry, with telephone contact visits one, four, and 28 weeks after entry and the week 48 visit. A physical exam and dental assessment was conducted at each clinic visit, and a history of adverse events collected. Dual Energy X-ray absorptiometry (DXA), hematology and chemistry panels were conducted at entry and weeks 24, 48, 72, 96 and 144. Lumbar spine and whole body (with head) BMD was measured using Hologic DXA scanners (QDR4500A, QDR4500W or Delphi A models).

The primary analysis compared changes from entry to 24 and 48 weeks in lumbar spine BMD between Groups 1A and 1B combined (both on alendronate for initial 48 weeks) vs. Group 2 (on placebo for 48 weeks). Study participants were unblinded after 96 weeks of follow-up (the primary completion date) but remained on study, off study treatment, for an additional 48 weeks.

Secondary laboratory outcomes listed in the protocol (bone marker turnover and Receptor Activator of Nuclear Factor Kappa-B Ligand/Osteoprotegerin (RANKL/OPG) Ratio) and central fat content, which required application for additional funding for laboratory testing, will not be performed and no results will be available.

ELIGIBILITY:
Inclusion Criteria (Version 2.0 of protocol):

* Documentation of HIV-1 infection
* HIV-infection acquired before puberty
* For participants receiving antiretroviral therapy, must have been on the same antiretroviral agents for at least 12 weeks prior to study entry and have a viral load less than 10,000 copies/mL. For participants not receiving antiretroviral therapy, must have not been on antiretroviral agents for at least 12 weeks prior to study entry and have no indication for therapy
* Lumbar spine DXA BMD z-score less than -1.5 or history of fragility fracture within the prior 12 months (regardless of DXA result).
* Available for routine dental exam and care every 6 months
* Demonstrated ability and willingness to swallow study medications
* Females of reproductive potential must have had a negative pregnancy test at screening and within 48 hours prior to study entry. They must also have agreed to avoid pregnancy while on the study and if engaging in sexual activity, use at least two forms of contraception.
* Parent or legal guardian able and willing to provide signed informed consent for children who could not provide consent for themselves.

Exclusion Criteria (Version 2.0 of protocol):

* Body weight more than 300 lbs.
* For female participants: if on Depo-Provera, they must have been on it for at least 1 year prior to study entry; if not on Depa-Provera, they must have not been on it for at least 1 year prior to study entry.
* Anticonvulsant therapy
* Proven growth hormone deficiency
* Use of growth hormone in the 12 months prior to entry
* Primary hyperparathyroidism
* Hypoparathyroidism
* Renal failure
* Cushing syndrome
* Active dental infection
* Dental or periodontal disease expected to require more than basic restorative care
* Pregnancy or lactation
* Esophageal or gastric ulcer, chronic nonsteroidal anti-inflammatory drug (NSAID) use, or aspirin use
* Tenofovir disoproxil fumarate (TDF): if on TDF, they must have been on it for at least 6 months prior to study entry; if not on TDF, they must have not been on it for at least 6 months prior to study entry.
* Hemoglobin less than 10 g/dL
* Any past pharmacologic treatment (except vitamin D and/or calcium supplementation) for low bone density
* Inability to stand or sit upright for at least 30 minutes
* Hypersensitivity to any component of alendronate
* Hypocalcemia (less than the lower limit of normal established by the local laboratory in which it was performed)
* Known abnormalities of the esophagus that delay esophageal emptying such as stricture or achalasia
* 25-OH vitamin D less than 10 ng/mL in combination with elevated intact PTH above the upper limit of normal for the local laboratory in which it was performed

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George K. Siberry, MD, Study Chair — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (10):
- United States (7):
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
- Brazil (2):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clay PG, Voss LE, Williams C, Daume EC. Valid treatment options for osteoporosis and osteopenia in HIV-infected persons. Ann Pharmacother. 2008 May;42(5):670-9. doi: 10.1345/aph.1K465. Epub 2008 Apr 15. PMID 18413693
- [Background] McComsey GA, Kendall MA, Tebas P, Swindells S, Hogg E, Alston-Smith B, Suckow C, Gopalakrishnan G, Benson C, Wohl DA. Alendronate with calcium and vitamin D supplementation is safe and effective for the treatment of decreased bone mineral density in HIV. AIDS. 2007 Nov 30;21(18):2473-82. doi: 10.1097/QAD.0b013e3282ef961d. PMID 18025884
- [Background] Stoch SA, Saag KG, Greenwald M, Sebba AI, Cohen S, Verbruggen N, Giezek H, West J, Schnitzer TJ. Once-weekly oral alendronate 70 mg in patients with glucocorticoid-induced bone loss: a 12-month randomized, placebo-controlled clinical trial. J Rheumatol. 2009 Aug;36(8):1705-14. doi: 10.3899/jrheum.081207. Epub 2009 Jun 1. PMID 19487264
- [Background] The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009).
- [Derived] Jacobson DL, Lindsey JC, Gordon C, Hazra R, Spiegel H, Ferreira F, Amaral FR, Pagano-Therrien J, Gaur A, George K, Benson J, Siberry GK. Alendronate Improves Bone Mineral Density in Children and Adolescents Perinatally Infected With Human Immunodeficiency Virus With Low Bone Mineral Density for Age. Clin Infect Dis. 2020 Aug 22;71(5):1281-1288. doi: 10.1093/cid/ciz957. PMID 31573608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-two (52) study participants were recruited between November 5, 2009 and March 27, 2014, at 10 study sites: 8 in the United States and 2 in Brazil.
Pre-assignment Details: Children and adolescents were randomly assigned to 3 treatment sequence groups. Two participants were enrolled, but because their baseline lumbar spine bone mineral density z-score was greater than -1.5 at their baseline visit, they never started study treatment and were taken off the study.
Groups:
- 1A: Alendronate/Alendronate: Participants received alendronate for 96 weeks
- 1B: Alendronate/Placebo: Participants received alendronate for 48 weeks followed by placebo for 48 weeks
- 2: Placebo/Alendronate: Participants received placebo for 48 weeks followed by alendronate for 48 weeks
Period: Weeks 0-48 (on Study Treatment)
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Started | 17 | 17 | 18
Completed | 15 (Completed 48 weeks) | 17 (Completed 48 weeks) | 18 (Completed 48 weeks)
Not Completed | 2 | 0 | 0
Not completed — Baseline lumbar spine > -1.5 | 2 | 0 | 0
Period: Weeks 48-96 (on Study Treatment)
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Started | 15 | 17 | 18
Completed | 15 | 16 | 17
Not Completed | 0 | 1 | 1
Not completed — Site Closure | 0 | 1 | 0
Not completed — Became a ward of the state | 0 | 0 | 1
Period: Weeks 96-144 (Off Study Treatment)
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Started | 15 | 16 | 17
Completed | 12 | 15 | 16
Not Completed | 3 | 1 | 1
Not completed — Site closure | 1 | 0 | 0
Not completed — Not able to attend clinic | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Includes participants who took at least one dose of study treatment (alendronate/placebo)
Groups:
- Total: Total of all reporting groups
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate | Total
Number analyzed (Participants) | 15 | 17 | 18 | 50
Age, Continuous [Median (Full Range); unit: years] | 16 [11 to 23] | 16 [12 to 23] | 16 [11 to 22] | 16 [11 to 23]
Age, Customized [Count of Participants; unit: Participants]
  11 - < 15 years | 7 | 4 | 6 | 17
  15 - < 19 years | 6 | 9 | 8 | 23
  >= 19 years | 2 | 4 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 10 | 11 | 13 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 3 | 3 | 1 | 7
  Black non-Hispanic | 2 | 4 | 1 | 7
  Hispanic (regardless of race) | 10 | 10 | 16 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 7 | 21
  Brazil | 9 | 9 | 11 | 29
Tanner stage [Count of Participants; unit: Participants] — Tanner stage represents the extent of physical development in children, adolescents and adults. It is based on external physical characteristics such as the size of breasts, genitals and pubic hair. Before puberty children are Tanner 1. Adults are Tanner 5. Study participants were classified as the most advanced stage of breasts and pubic hair (females) and genitals and pubic hair (males).
  Participants
    1 | 1 | 0 | 2 | 3
    2 | 3 | 2 | 2 | 7
    3 | 5 | 1 | 2 | 8
    4 | 1 | 8 | 6 | 15
    5 | 5 | 6 | 6 | 17
Smoker [Count of Participants; unit: Participants]
  Yes | 0 | 2 | 1 | 3
  No | 15 | 15 | 17 | 47
Bone age [Median (Full Range); unit: years] — Population: Bone age estimates maturity of a child's skeletal system. It was assessed by taking an X-ray of the left wrist, hand, and fingers. the X-ray was compared with images in a standard atlas of bone development, based on data from large numbers of other kids of the same gender and age. One participant did not have bone age measured at entry.
  years
    number analyzed (Participants) | 15 | 16 | 18 | 49
    (all) | 14 [10 to 22] | 16 [11 to 23] | 15 [11 to 21] | 15 [10 to 23]
Use of tenofovir [Count of Participants; unit: Participants] — Tenofovir disoproxil is a drug used to treat HIV
  Participants
    Yes | 7 | 7 | 9 | 23
    No | 8 | 10 | 9 | 27
CDC HIV disease category [Count of Participants; unit: Participants] — Severity of HIV disease was classified using the Centers for Disease Control (CDC) 1993 Revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults (https://www.cdc.gov/mmwr/preview/mmwrhtml/00018871.htm). Disease category C/3 is the most advanced.
  Participants
    A/1 | 0 | 1 | 3 | 4
    B/2 | 2 | 0 | 6 | 8
    C/3 | 13 | 16 | 9 | 38
HIV-1 RNA (copies/ml) [Count of Participants; unit: Participants]
  <= 400 | 10 | 16 | 15 | 41
  >400 | 5 | 1 | 3 | 9
CD4 cell count (cells/mm^3) [Count of Participants; unit: Participants]
  200 - <500 | 3 | 3 | 2 | 8
  500 - < 1000 | 10 | 10 | 10 | 30
  >= 1000 | 2 | 4 | 6 | 12
25-OH Vitamin D (ng/mL) [Count of Participants; unit: Participants]
  10 - < 20 | 1 | 5 | 0 | 6
  20 - < 30 | 7 | 8 | 6 | 21
  >= 30 | 7 | 4 | 12 | 23
Lumbar spine BMD (g/cm^2) [Median (Full Range); unit: g/cm^2] | 0.64 [0.47 to 0.93] | 0.73 [0.50 to 0.89] | 0.66 [0.50 to 0.88] | 0.70 [0.47 to 0.93]
Whole body (with head) BMD (g/cm^2) [Median (Full Range); unit: g/cm^2] — Population: Whole body (with head) BMD was missing at entry for some participants because of software problems with the DXA machines.
  g/cm^2
    number analyzed (Participants) | 14 | 16 | 16 | 46
    (all) | 0.87 [0.68 to 1.05] | 0.91 [0.62 to 1.08] | 0.86 [0.69 to 1.08] | 0.87 [0.62 to 1.08]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Weeks 24 and 48 in Lumbar Spine BMD
Description: Percent change was calculated as (measurement at time T - measurement at baseline)/measurement at baseline * 100%. Results for Groups 1A and 1B combined as both were on alendronate for the first 48 weeks.
Time Frame: Weeks 0, 24 and 48
Population: Includes all participants who started study treatment
Measure: Median (95% Confidence Interval); unit: Percent change from baseline
Groups:
- 1: Alendronate: Participants received alendronate for 48 weeks
- 2: Placebo: Participants received placebo for 48 weeks
Arm/Group | 1: Alendronate | 2: Placebo
Number analyzed (Participants) | 32 | 18
Percent change from baseline
  Week 24 | 14.4 [8.8 to 19.4] | 5.5 [1.2 to 7.6]
  Week 48 | 15.9 [9.2 to 25.3] | 7.1 [4.9 to 8.9]
Statistical Analysis 1: Comparison: 1: Alendronate vs 2: Placebo; Comparison of percent change from baseline to week 24; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: 1: Alendronate vs 2: Placebo; Comparison of percent change from baseline to week 48; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons

2. Primary Outcome: Percentage of Participants Developing New Signs, Symptoms, Hematology or Chemistry Laboratory Values Greater Than or Equal to Grade 3 or New Cases of Jaw Osteonecrosis, Atrial Fibrillation, or Non-healing Fractures
Description: Signs, symptoms, and laboratory values were graded using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0 (December 2004). Results for Groups 1A and 1B were combined as both were on alendronate for the first 48 weeks.
Time Frame: Week 0 to 48
Population: All participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Alendronate | 2: Placebo
Number analyzed (Participants) | 32 | 18
Participants | 5 | 2
Statistical Analysis 1: Comparison: 1: Alendronate vs 2: Placebo; Comparison of percentage of participants experiencing primary safety outcome; Test type: Superiority or Other; p > 0.99, Fisher Exact — Not adjusted for multiple comparisons

3. Secondary Outcome: Percent Change From Baseline to Weeks 24 and 48 in Whole Body (With Head) BMD
Description: Percent change was calculated as (measurement at time T - measurement at baseline)/measurement at baseline * 100%. Results for Groups 1A and 1B were combined as both were on alendronate for the first 48 weeks.
Time Frame: Weeks 0, 24 and 48
Population: Participants who started treatment and had Whole Body (with head) BMD available at week 0
Measure: Median (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 1: Alendronate | 2: Placebo
Number analyzed (Participants) | 30 | 16
Percent change from baseline
  Week 24 | 5.5 [3.7 to 8.1] | 0.3 [-0.5 to 3.6]
  Week 48: number analyzed (Participants) | 29 | 16
  Week 48 | 10.7 [6.0 to 16.2] | 5.2 [1.6 to 8.5]

4. Secondary Outcome: Percent Change From Baseline to Week 96 in Lumbar Spine BMD
Description: Percent change was calculated as (measurement at week 96 - measurement at baseline)/measurement at baseline * 100%. Includes Groups 1A and 1B only.
Time Frame: Weeks 0 and 96
Population: Includes all participants who started study treatment and had measurements available at weeks 0 and 96
Measure: Median (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo
Number analyzed (Participants) | 14 | 16
Percent change from baseline | 24.9 [11.1 to 69.8] | 14.8 [11.4 to 32.6]

5. Secondary Outcome: Percent Change From Baseline to Week 96 in Whole Body (With Head) BMD
Description: as for outcome 4
Time Frame: Weeks 0 and 96
Population: Includes all participants who started study treatment and had measurements available at weeks 0 and 96
Measure: Median (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo
Number analyzed (Participants) | 12 | 14
Percent change from baseline | 19.6 [7.7 to 30.4] | 10.3 [5.1 to 24.9]

6. Secondary Outcome: Safety as Measured by the Incidence of New Signs, Symptoms, Hematology or Chemistry Laboratory Values Greater Than or Equal to Grade 3 or New Cases of Jaw Osteonecrosis, Atrial Fibrillation, or Non-healing Fractures
Description: Signs, symptoms, and laboratory values were graded using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0 (December 2004).
Time Frame: Weeks 0 to 144
Population: All participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 15 | 17 | 18
Participants
  Week 0 to 48 | 2 | 3 | 2
  Week 48 to 96 | 1 | 3 | 2
  Week 96 to 144: number analyzed (Participants) | 15 | 16 | 17
  Week 96 to 144 | 3 | 4 | 3

7. Secondary Outcome: Effect of Other Known Bone Mineral Determinants (Age, Gender, Race/Ethnicity, Steroid Use, Depo-Provera, Tenofovir, Pubertal Stage, Bone Age, Vitamin D Status) and Inflammatory Cytokine Levels on Changes in Lumbar Spine BMD
Description: A slope was fit for each participant to their percent change [(measurement at time T - measurement at baseline)/measurement at baseline)*100%] in lumbar spine BMD from baseline. Results represent average changes in lumbar spine BMD over one year. Results are summarized for age, gender, ethnicity, tenofovir use, Tanner stage, bone age and vitamin D level. Only one participant was on steroids and none were using Dep-Provera. Inflammatory cytokine levels were not assayed. Results were combined for Groups 1A and 1B as both were on alendronate for the first 48 weeks.
Time Frame: Weeks 0, 24 and 48
Population: Participants who started study treatment
Measure: Mean (95% Confidence Interval); unit: percentage of baseline
Arm/Group | 1: Alendronate | 2: Placebo
Number analyzed (Participants) | 32 | 18
percentage of baseline
  Male: number analyzed (Participants) | 21 | 13
  Male | 20.3 [13.0 to 27.6] | 6.8 [4.7 to 8.8]
  Female: number analyzed (Participants) | 11 | 5
  Female | 25.4 [13.3 to 37.5] | 9.4 [-0.1 to 18.9]
  Non-hispanic: number analyzed (Participants) | 12 | 2
  Non-hispanic | 19.4 [7.6 to 31.1] | 4.8 [-1.4 to 11.1]
  Hispanic: number analyzed (Participants) | 20 | 16
  Hispanic | 23.6 [16.3 to 31.0] | 7.8 [5.2 to 10.5]
  11 - < 15 years: number analyzed (Participants) | 11 | 6
  11 - < 15 years | 37.1 [27.7 to 46.5] | 10.6 [5.6 to 15.7]
  15 - < 19 years: number analyzed (Participants) | 15 | 8
  15 - < 19 years | 16.5 [9.6 to 23.4] | 8.0 [5.8 to 10.1]
  >= 19 years: number analyzed (Participants) | 6 | 4
  >= 19 years | 8.1 [-0.7 to 16.9] | 1.9 [-4.4 to 8.2]
  On Tenofovir: number analyzed (Participants) | 14 | 9
  On Tenofovir | 24.8 [15.1 to 34.5] | 6.8 [3.6 to 10.0]
  Not on Tenofovir: number analyzed (Participants) | 18 | 9
  Not on Tenofovir | 19.9 [11.6 to 28.2] | 8.2 [3.9 to 12.5]
  25-OH Vit D<30 ng/ml: number analyzed (Participants) | 21 | 6
  25-OH Vit D<30 ng/ml | 22.0 [13.5 to 30.4] | 6.8 [1.9 to 11.7]
  25-0H Vit D>=30 ng/ml: number analyzed (Participants) | 11 | 12
  25-0H Vit D>=30 ng/ml | 22.1 [13.5 to 30.8] | 7.8 [4.6 to 11.0]
  Bone age < 15 years: number analyzed (Participants) | 12 | 9
  Bone age < 15 years | 36.0 [28.1 to 43.9] | 10.0 [6.9 to 13.0]
  Bone age>=15 years: number analyzed (Participants) | 19 | 9
  Bone age>=15 years | 11.3 [7.6 to 15.1] | 5.0 [1.6 to 8.4]
  Tanner stage <= 3: number analyzed (Participants) | 12 | 6
  Tanner stage <= 3 | 33.0 [22.7 to 43.3] | 10.6 [5.6 to 15.7]
  Tanner stage >= 4: number analyzed (Participants) | 20 | 12
  Tanner stage >= 4 | 15.4 [9.2 to 21.6] | 5.9 [3.3 to 8.6]

8. Secondary Outcome: Effect of Other Known Bone Mineral Determinants (Age, Gender, Race/Ethnicity, Steroid Use, Depo-Provera, Tenofovir, Pubertal Stage, Bone Age, Vitamin D Status) and Inflammatory Cytokine Levels on Changes in Whole Body (With Head) BMD.
Description: A slope was fit for each participant to their percent change [(measurement at time T - measurement at baseline)/measurement at baseline)*100%] in whole body (with head) BMD from baseline. Results represent average changes in whole body (with head) BMD over one year. Results are summarized for age, gender, ethnicity, tenofovir use, Tanner stage, bone age and vitamin D level. Only one participant was on steroids and none were using Dep-Provera. Inflammatory cytokine levels were not assayed. Results were combined for Groups 1A and 1B as both were on alendronate for the first 48 weeks.
Time Frame: Weeks 0, 24 and 48
Population: Participants who started study treatment and had Whole Body (with head) available at week 0
Measure: Mean (95% Confidence Interval); unit: percentage of baseline
Arm/Group | 1: Alendronate | 2: Placebo
Number analyzed (Participants) | 30 | 16
percentage of baseline
  Male: number analyzed (Participants) | 20 | 11
  Male | 11.4 [7.4 to 15.3] | 4.1 [1.1 to 7.1]
  Female: number analyzed (Participants) | 10 | 5
  Female | 14.0 [6.0 to 22.0] | 8.2 [1.6 to 14.7]
  Non-Hispanic: number analyzed (Participants) | 12 | 2
  Non-Hispanic | 9.8 [2.7 to 17.0] | 0.3 [-4.4 to 4.9]
  Hispanic: number analyzed (Participants) | 18 | 14
  Hispanic | 13.9 [10.0 to 17.7] | 6.1 [3.3 to 8.9]
  11 - < 15 years: number analyzed (Participants) | 10 | 6
  11 - < 15 years | 19.2 [12.9 to 25.5] | 8.0 [2.9 to 13.2]
  15 - < 19 years: number analyzed (Participants) | 14 | 6
  15 - < 19 years | 10.5 [6.1 to 14.9] | 6.5 [3.0 to 10.0]
  >= 19 years: number analyzed (Participants) | 6 | 4
  >= 19 years | 4.7 [-2.0 to 11.4] | -0.3 [-3.8 to 3.2]
  On tenofovir: number analyzed (Participants) | 12 | 9
  On tenofovir | 13.2 [7.6 to 18.8] | 5.0 [1.5 to 8.6]
  Not on tenofovir: number analyzed (Participants) | 18 | 7
  Not on tenofovir | 11.6 [6.7 to 16.5] | 5.8 [0.5 to 11.2]
  25-0H Vit D<30 ng/ml: number analyzed (Participants) | 19 | 5
  25-0H Vit D<30 ng/ml | 10.6 [5.6 to 15.6] | 5.8 [-2.7 to 14.3]
  25-0H Vit D>=30 ng/ml: number analyzed (Participants) | 11 | 11
  25-0H Vit D>=30 ng/ml | 15.1 [10.6 to 19.5] | 5.2 [2.3 to 8.0]
  Bone age < 15 years: number analyzed (Participants) | 10 | 8
  Bone age < 15 years | 19.0 [14.7 to 23.3] | 8.4 [4.7 to 12.1]
  Bone age >=15 years: number analyzed (Participants) | 19 | 8
  Bone age >=15 years | 7.7 [4.1 to 11.2] | 2.3 [-0.6 to 5.2]
  Tanner stage <= 3: number analyzed (Participants) | 10 | 6
  Tanner stage <= 3 | 18.0 [10.5 to 25.5] | 8.0 [2.9 to 13.2]
  Tanner stage >= 4: number analyzed (Participants) | 20 | 10
  Tanner stage >= 4 | 9.4 [5.9 to 12.8] | 3.8 [0.6 to 7.0]

9. Secondary Outcome: Percent Change From Week 48 to Week 96 (Group 1B), Week 48 to Week 144 (Group 1B), and Week 96 to 144 (Group 2) in Lumbar Spine BMD
Description: Percent change was calculated as (measurement at time T2 - measurement at time T1)/measurement at Time T1 * 100%.
Time Frame: Weeks 48, 96 and 144
Population: All participants who started study treatment and had measurements available at the two time points of interest
Measure: Median (95% Confidence Interval); unit: Percent change
Groups:
- 1B: Alendronate/Placebo (48 Week Change); 1B: Alendronate/Placebo (96 Week Change): Participants received alendronate for 48 weeks followed by placebo for 48 weeks.
- 2: Placebo/Alendronate (48 Week Change): Participants received placebo for 48 weeks followed by alendronate for 48 weeks
Arm/Group | 1B: Alendronate/Placebo (48 Week Change) | 2: Placebo/Alendronate (48 Week Change) | 1B: Alendronate/Placebo (96 Week Change)
Number analyzed (Participants) | 15 | 15 | 15
Percent change | 0.9 [-1.1 to 6.4] | 2.0 [-0.6 to 4.6] | 1.7 [-1.0 to 6.1]

10. Secondary Outcome: Percent Change From Week 48 to Week 96 (Group 1B), Week 48 to Week 144 (Group 1B), and Week 96 to 144 (Group 2) in Whole Body (With Head) BMD
Description: Percent change was calculated as (measurement at time T2 - measurement at time T2)/measurement at time T1 * 100%.
Time Frame: Weeks 48, 96 and 144
Population: All participants who started study treatment and had measurements available at both time points.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | 1B: Alendronate/Placebo (48 Week Change) | 2: Placebo/Alendronate (48 Week Change) | 1B: Alendronate/Placebo (96 Week Change)
Number analyzed (Participants) | 15 | 13 | 15
Percent change | 0.8 [-1.9 to 3.1] | 0.5 [-0.4 to 2.1] | 0.9 [0.0 to 5.9]

11. Secondary Outcome: Change From Baseline to Week 48 in Bone Marker Turnover
Description: Outcome measure required additional funding for laboratory testing which was not available, so this outcome is not reported.
Time Frame: Weeks 0 and 48
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Correlation of Changes in Bone Marker Turnover With Changes in Lumbar Spine and Whole Body (With Head) BMD
Description: as for outcome 11
Time Frame: Weeks 0 and 48
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline to Week 48 in Receptor Activator of Nuclear Factor Kappa-B Ligand/Osteoprotegerin (RANKL/OPG) Ratio
Description: as for outcome 11
Time Frame: Weeks 0 and 48
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Correlation of Changes in RANKL/OPG Ratio With Changes in Lumbar Spine and Whole Body (With Head) BMD
Description: as for outcome 11
Time Frame: Weeks 0 and 48
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline to Week 48 in Central Fat Content
Description: as for outcome 11
Time Frame: Weeks 0 and 48
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Correlation of Changes in Central Fat Content With Changes in Lumbar Spine and Whole Body (With Head) BMD
Description: as for outcome 11
Time Frame: Weeks 0 and 48
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Percent of Participants With HIV-1 RNA <= 400 Copies/ml
Description: Percent calculated as number of participants with HIV-1 RNA <= 400 copies/ml relative to the number of participants with HIV-1 RNA measured at that time point.
Time Frame: Weeks 0, 48, 96 and 144
Population: Participants who started study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 15 | 17 | 18
Participants
  Week 0 | 10 | 16 | 15
  Week 48: number analyzed (Participants) | 15 | 17 | 16
  Week 48 | 10 | 16 | 14
  Week 96: number analyzed (Participants) | 14 | 15 | 17
  Week 96 | 12 | 12 | 13
  Week 144: number analyzed (Participants) | 12 | 14 | 16
  Week 144 | 10 | 10 | 10

18. Secondary Outcome: Change in CD4 Percent From Baseline
Description: Change in percentage of lymphocytes that are CD4 cells calculated as measurement at each time point minus baseline measurement
Time Frame: Weeks 0, 48, 96 and 144
Population: Participants who started study treatment and had CD4 percent available at week 0.
Measure: Median (95% Confidence Interval); unit: percent of lymphocytes that are CD4 cell
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 15 | 17 | 18
percent of lymphocytes that are CD4 cell
  Week 48 - Week 0: number analyzed (Participants) | 15 | 17 | 17
  Week 48 - Week 0 | 0 [-3 to 4] | 1 [-2 to 3] | 1 [-2 to 4]
  Week 96 - Week 0: number analyzed (Participants) | 14 | 15 | 17
  Week 96 - Week 0 | 0 [-5 to 4] | -1 [-3 to 3] | 2 [-4 to 3]
  Week 144 - Week 0: number analyzed (Participants) | 12 | 14 | 16
  Week 144 - Week 0 | 1 [-9 to 4] | -1 [-3 to 4] | -4 [-5 to 8]

19. Secondary Outcome: Change in Centers for Disease Control (CDC) HIV Disease Category
Description: Percentage of participants advancing in CDC HIV disease category from baseline throughout study follow-up
Time Frame: Weeks 144
Population: Participants who started study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 15 | 17 | 18
Participants
  Week 0 to 48 | 1 | 0 | 0
  Week 48 to 96 | 0 | 1 | 0
  Week 96 to 144: number analyzed (Participants) | 15 | 16 | 17
  Week 96 to 144 | 0 | 0 | 0

20. Secondary Outcome: Percent of Participants With Detectable Urinary Alendronate
Description: as for outcome 11
Time Frame: Weeks 48, 96 and 144
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to end of follow-up (144 weeks)
Description: Expedited adverse event (EAE) reporting followed the DAIDS EAE Manual under the SAE Reporting Category and including fetal losses. Events were graded (1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death) according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Clarification Aug 2009. Reports are summarized by randomized arm for consistency with outcomes and because effects of alendronate can continue for months after stopping the drug.
Groups:
- 1A: Alendronate/Alendronate: Participants received alendronate for 48 weeks
Arm/Group | 1A: Alendronate/Alendronate | 1B: Alendronate/Placebo | 2: Placebo/Alendronate
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/17 | 3/18
Other Adverse Events (participants affected / at risk) | 15/15 | 17/17 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1A: Alendronate/Alendronate (N=15) | 1B: Alendronate/Placebo (N=17) | 2: Placebo/Alendronate (N=18)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1A: Alendronate/Alendronate (N=15) | 1B: Alendronate/Placebo (N=17) | 2: Placebo/Alendronate (N=18)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 1 | 1
Myopia (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Lip blister (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 1
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Tooth discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 7
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Chest pain (General disorders) | 3 | 1 | 4
Fatigue (General disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 1 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 2 | 2
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 2
Flea infestation (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 1
Gingivitis (Infections and infestations) | 1 | 4 | 3
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 3
Oral herpes (Infections and infestations) | 2 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 2
Otitis media (Infections and infestations) | 1 | 3 | 2
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Scarlet fever (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Sinusitis bacterial (Infections and infestations) | 2 | 2 | 3
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 2 | 2 | 1
Tonsillitis (Infections and infestations) | 2 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 3
Aspartate aminotransferase (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase abnormal (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 6 | 2 | 4
Blood bicarbonate decreased (Investigations) | 2 | 4 | 4
Blood bilirubin increased (Investigations) | 2 | 4 | 6
Blood calcium decreased (Investigations) | 0 | 0 | 1
Blood calcium increased (Investigations) | 3 | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 2 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 4
Blood glucose decreased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 2
Blood pH decreased (Investigations) | 2 | 1 | 2
Blood phosphorus decreased (Investigations) | 4 | 3 | 4
Blood potassium decreased (Investigations) | 0 | 1 | 2
Blood sodium decreased (Investigations) | 5 | 2 | 7
Blood sodium increased (Investigations) | 0 | 2 | 2
Blood uric acid increased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 2
Heart rate irregular (Investigations) | 1 | 0 | 0
Lipase abnormal (Investigations) | 1 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 2 | 2 | 6
Platelet count decreased (Investigations) | 2 | 2 | 1
Prothrombin time abnormal (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 2
Body fat disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 3
Headache (Nervous system disorders) | 3 | 2 | 2
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 2
Seizure (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Abortion early (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 2 | 1
Substance abuse (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal tubular dysfunction (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights